CLINICAL TRIAL: NCT06737133
Title: Early Management of Fracture Nose in Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yara Asem Althany Mohamed, Physician, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-11-07MS
Record Dates: First submitted 2024-11-25; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Fracture Nose
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery — Rhinoplasty

SUMMARY:
Introduction:

Nasal fractures are common components of the facial skeleton injuries. Nasal bone fractures are the most common type of facial fracture (1), and the third most common fracture of the human skeleton (2).

Nasal fractures are frequently associated with cartilaginous and soft tissue injuries. The incidence of post- traumatic nasal deformity, if left untreated, varies from 14% to 50% (3).The management of nasal injuries since Maliniac's description of the management of nasal fractures in 1947 has seen several variations (3) .

The functional and cosmetic problems arising may sometimes necessitate intricate surgical procedures to restore the anatomy. Due to constraints of resources and the range of services provided, these injuries are typically managed . Most commonly, nasal bone fractures are sustained in fights (34%), accidents (28%), and sports (23%). A 2009 study of 236 patients with facial fractures incurred while playing sports determined that fractures of the nasal bone were most common (4) . In children, nasal fractures are most commonly due to falls. In a study of 100 children with traumatic nasal deformity, Liu et al determined that such injuries were most often the result of sports-related trauma (28%), with accidental trauma (21%), interpersonal violence (10%), motor vehicle collisions (6%), and alcohol- related trauma (2%) being the next most common reasons for injury (5) . The possibility of child abuse should be considered in every child presenting with a nasal fracture The prognosis of nasal bone fracture is depend on: If NBFs are treated within correct time parameters, patients should anticipate a successful healing and proper nasal alignment. Communication between the surgeon, ENT physician, and primary care physician or emergency physician is crucial to the treatment plan (6). The greatest complications from reduction are malunion and cosmetic concerns. Incidence of complications is highest in bilateral fractures, comminuted fractures, and fractures with severe nasal septum deviation (7).

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from since birth to 12 years old
* Isolated nasal fracture
* Presented from time of trauma up to 5 days

Exclusion Criteria:

* Multiple facial fractures
* Age more than 12 years old
* Systemic diseases
* Any hematological disorders

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Measure of the outer framework of the nose after trauma | One year and 3 months
  Early correction of nasal fractures to preserve the outer framework of the nose after trauma achieving the best result aiming to minimize rhinoplasty further on ,measuring the nasal bone length pre and postoperative